CLINICAL TRIAL: NCT05035667
Title: Social Media Use in Advanced Cancer: Patient Considerations of Social Media Account Management After Death
Brief Title: Patient Considerations of Social Media Account Management After Death
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1171; NCI-2021-04176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1171 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-21; First posted 2021-09-05 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid System Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaires): Patients complete questionnaires over 30 minutes about level of anxiety and social media use and management.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines how supportive care clinic patients have made decisions or had discussions about how their caregivers or family should manage their social media account(s) after death. Collecting information on the use of social media and preferences will allow for a better understanding of patient's needs in the dying process and may identify populations in need of education, identify a possible source of anxiety and stress, and allow for an informed discussion of digital legacy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Identify the proportion of patients with advanced cancer in the supportive cancer clinic who have had discussions regarding their social media account (e.g. Facebook, Twitter, Instagram) management after death.

SECONDARY OBJECTIVE:

I. Identify the proportion of social media participation among advanced cancer patients seen in the supportive care clinic.

II. Evaluate the baseline awareness advanced cancer patients seen in the supportive care clinic have regarding how their Facebook account may be managed after death.

III. Evaluate affect changes and distress as a result from the conversation regarding their social media account management after death.

IV. Evaluate if discussion of social media account management among patients with advanced cancer in the supportive cancer clinic will increase their awareness of and motivation to address their social media account management options.

OUTLINE:

Patients complete questionnaires over 30 minutes about level of anxiety and social media use and management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 1 follow-up visit to the outpatient Supportive Care Clinic at MDACC
* Patients with any type of advanced cancer
* Patients aged 18 years or older
* Patients who have used social media
* Patients able to read and write in English

Exclusion Criteria:

* Delirium as diagnosed by treating Supportive Care Center (SCC) physician or Memorial Delirium Assessment Scale (MDAS) score >= 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer attending outpatient Supportive Care Clinic at M D Anderson Cancer Center (MDACC)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with advanced cancer in the supportive cancer clinic who have had discussions regarding their social media account | through study completion, an average of 1 year
  Will be measured by Question 10 in the survey: "I have had conversations with my family or friends regarding how I would like any of my social media accounts managed after death", which contains five options: Strongly Disagree, Disagree, Neither Agree or Disagree, Agree, or Strongly Agree. The results will be dichotomized into either "Strongly Agree/Agree" or "Neither Agree or Disagree/ Disagree/Strongly Disagree". A two-sided 95% confidence interval will extend a maximum of 0.063 from the proportion of main interest.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline M Tschanz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org